CLINICAL TRIAL: NCT04734223
Title: Correlation of Neuroimaging Findings With Clinical Presentation and Laboratory Data in Patients With COVID-19: A Single Center Study
Brief Title: Neuroimaging Findings in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyhmus Kavak, MD, Radiologist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 09.25.2020/587
Record Dates: First submitted 2021-01-29; First posted 2021-02-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Neuroimaging; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: The first group consisted of 46 patients whose neuroimaging findings demonstrated acute/subacute infarction, bleeding, encephalitis, and venous sinus thrombosis
  Interventions: Diagnostic Test: Neuroimaging Findings in Patients With COVID-19
- Group 2: The 2nd group (N=390) was obtained by subtracting the 1st group from all cases.
  Interventions: Diagnostic Test: Neuroimaging Findings in Patients With COVID-19
- Group 3: The third group (N = 189) consisted of patients of the first group and patients with chronic ischemic changes observed in neuroimaging
  Interventions: Diagnostic Test: Neuroimaging Findings in Patients With COVID-19
- Group 4: The 4th group (N=247) was obtained by subtracting the 3rd group from all cases.
  Interventions: Diagnostic Test: Neuroimaging Findings in Patients With COVID-19

INTERVENTIONS:
Diagnostic Test: Neuroimaging Findings in Patients With COVID-19 — MR and BT Imaging

SUMMARY:
This study aimed to discuss the neuroimaging findings and indications, epidemiological data, laboratory values, and the relationship of these variables with mortality in patients with COVID-19.

DETAILED DESCRIPTION:
COVID-19 can present as neurological symptoms such as anosmia, headache, taste perversion, dizziness, syncope, and altered state of consciousness. It has been reported in previous studies that thromboembolic ischemic and hemorrhagic strokes associated with COVID-19 have been observed in the early period. It has been suggested that conditions characterized by neurological sequelae, such as encephalitis and encephalopathy, ataxic seizures, Guillain-Barré syndrome (GBS), demyelinating diseases, and neuromuscular disorders may occur in the longer term.In the present study, the investigators aimed to reveal the findings of neuroimaging analyses performed in patients followed up with a diagnosis of COVID-19 who had neurological symptoms, discuss the relationship of these findings with laboratory and epidemiological data, and emphasize that CNS involvement in these patients should not be overlooked. In this study, 436 patients with COVID-19 who underwent at least one neuroimaging procedure during April 2020-December 2020 due to neurological symptoms and whose diagnosis was confirmed by reverse transcriptase-polymerase chain reaction test were included. Although computed tomography was predominantly used for imaging, magnetic resonance imaging was also used when necessary. The patients were grouped based on imaging findings, and statistical evaluations were made between the groups.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 RT-PCR positivity-
* older than 18 years old

Exclusion Criteria:

* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects more than 18 years old and who are followed up and treated with the diagnosis of COVID-19 in Sağlık Bilimleri Üniversitesi Gazi Yaşargil Training and Research Hospital will be included.
Sampling Method: Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of acute thromboembolism in COVID-19 patients undergoing neuroimaging | Between April and December 2020
  Acute thromboembolic events are common in COVID-19 subjects undergoing neuroimaging, potentially due to an increased procoagulant process.

CONTACTS AND LOCATIONS:
Overall Officials: ŞEYHMUS KAVAK, MD, Principal Investigator — SAGLIK BİLİMLERİ ÜNİVERSİTESİ TRAINING AND RESEARCH HOSPITAL H
Locations (1):
- Sağlik Bilimleri Üniversitesi Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided